CLINICAL TRIAL: NCT01791257
Title: MicroRNA Expression in Cerebrospinal Fluid From Patients Suffering Subarachnoid Hemorrhage With and Without Delayed Cerebral Ischemia
Brief Title: MicroRNA Diagnostics in Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Søren Bache Larsen, MD, MD, Rigshospitalet, Denmark
Other Study IDs: MicroRNA in SAH
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Subarachnoid Hemorrhage
Keywords: delayed; cerebral; ischemia; microrna; cerebrospinal fluid; subarachnoid; hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage; Ischemia; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Group 1+2: Cerebrospinal fluid 1-2 ml a day for 8 days drawn in each patient from external ventricular drain Gropu 3: Cerebrospinal fluid 2 ml drawn from patients undergoing spinal anesthesia before injection of local anesthetic.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- SAH with DCI: After 21 days from ictus the patients with subarachnoid hemorrhage are stratified to group 1 or 2 depending on their development of delayed cerebral ischemia.
- SAH without DCI: After 21 days from ictus the patients with subarachnoid hemorrhage are stratified to group 1 or 2 depending on their development of delayed cerebral ischemia.
- Neurological healthy controls: 12 patients (ASA 1) undergoing spinal anesthesia for orthopedic surgery have 2 ml of cerebrospinal fluid drawn preceding injection of local analgetic.

SUMMARY:
The purpose of this study is to compare the profile of microRNA in cerebrospinal fluid from patients suffering subarachnoid hemorrhage with and without delayed cerebral ischemia.

DETAILED DESCRIPTION:
In this study of patients suffering an aneurysmal subarachnoid hemorrhage (SAH) we would like to investigate the pathophysiological mechanisms that lead to the phenomenon delayed cerebral ischemia (DCI).

We will accomplish this through analyzing the profile of microRNA expression in the cerebrospinal fluid of SAH patients treated with extraventricular drainage.

At first we wish to compare the expression of 376 specific microRNA between 12 patients developing DCI (group 1) and 12 patients without DCI (group 2) in cerebrospinal fluid drawn on day 5 after ictus.

Secondly specific microRNAs of interest in which the expression differs between group 1 and 2 are analyzed daily to investigate the dynamic changes in expression and compared to the clinical course.

Should we find no differently expressed specific microRNAs we will compare the expression of microRNA in group 1+2 with group 3.

In addition, some of the patients as part of another clinical trial (NCT01447095

) will have established invasive neuromonitoring including microdialysis. It is our intention to develop a method for analyzing microRNA in this microdialysate.

DCI as defined by Vergouwen et al in Stroke 2010;41(10):2391-2395:

"The occurrence of focal neurological impairment (such as hemiparesis, aphasia, apraxia, hemianopia, or neglect), or a decrease of at least 2 points on the Glasgow Coma Scale (either on the total score or on one of its individual components [eye, motor on either side, verbal]). This should last for at least 1 hour, is not apparent immediately after aneurysm occlusion, and cannot be attributed to other causes by means of clinical assessment, CT or MRI scanning of the brain, and appropriate laboratory studies."

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the neurointensive care unit with aneurismal subarachnoid hemorrhage
* External ventricular drainage with 5 days of ictus
* Age > 18 years

Exclusion Criteria:

* Glasgow Coma Score (GCS) continuously < 7 during the first 5 days following ictus
* A known and proven complication (rebleeding, clip/coil complication, cardiopulmonal complication requiring full sedation, ventriculitis e.g.) leads to a GCS < 7 thereby preventing the detection of DCI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1+2: Patients admitted to Neurointensive Department in Rigshospitalet. Group 3: Patients undergoing spinal anesthesia for orthopedic surgery in Bispebjerg Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Delayed Cerebral Ischemia - Clean groups | 21 days
  Delayed Cerebral Ischemia as defined by Vergouwen et al in Stroke 2010;41(10):2391-2395.
  We found confirmation/exclusion of DCI difficult in a few patients. To minimize error, two clinicians reviewed all clinical, biochemical and radiological data, obtained 3 weeks from ictus, and independently assessed if any clinical deterioration fulfilled the criteria of delayed cerebral ischemia. Furthermore, included patients were categorized as "definitely DCI", "probably DCI", "probably not DCI" or "definitely not DCI".
  Therefore we decided to modify our primary outcome measure in this case-control study to compare "definitely DCI" vs. "definitely not DCI".

SECONDARY OUTCOMES:
Early brain injury: Comparison of microRNA profiles with clinical neurology following occlusion of the aneurysm | Assessed at the first wake-up call following clip or coil
  Comparison of 667 specific microRNAs in CSF at day 5 after ictus between two groups of SAH-patients depending on their clinical neurology at the first wake-up call following occlusion of the aneurysm:
  1. GCS 3-12 and/or (paresis (degree 4) of at least one extremity or aphasia)
  2. GCS 13-15 and no or only small and mild focal deficit
Association of microRNA-profile with 3 month outcome | Follow up examination at 3 month or as close to this
  Comparison of 667 specific microRNAs in CSF at day 5 after ictus between two groups of SAH-patients depending on their mRS at 3 month follow-up in groups:
  1. mRS = 3-6
  2. mRS = 0-2
Delayed Cerebral Ischemia as defined by Vergouwen et al in Stroke 2010;41(10):2391-2395. Large groups. | 21 days following ictus
  Delayed Cerebral Ischemia as defined by Vergouwen et al in Stroke 2010;41(10):2391-2395.
  In contrast to our primary outcome measure, these groups will include patients where DCI was difficult to exclude or confirm.
  Thereby we wish to compare "definitely DCI" and "probably DCI" vs. "probably not DCI" and "definetly not DCI". This would enable comparison between larger groups though less clean.
Relation of microRNA profile to cerebral infarction as defined by Vergouwen et al in Stroke 2010;41(10):2391-2395. | Following a blinded description of CT-scans
  The presence of cerebral infarction on CT or MR scan of the brain within 6 weeks after SAH, or on the latest CT or MR scan made before death within 6 weeks, or proven at autopsy, not present on the CT or MR scan between 24 and 48 hours after early aneurysm occlusion, and not attributable to other causes such as surgical clipping or endovascular treatment. Hypodensities on CT imaging resulting from ventricular catheter or intraparenchymal hematoma should not be regarded as cerebral infarctions from DCI.
Relation of microRNA profile to the regional area of cerebral injury | Following a blinded description of CT-scans
  As microRNAs seem to be specific for different areas of the brain our screening might tell us which area has sustained injury and which has not. This study will not include two groups as the secondary outcome measures above.

CONTACTS AND LOCATIONS:
Overall Officials: Søren B Larsen, MD, Principal Investigator — Rigshopsitalet, Denmark; Kirsten Møller, DMSci, Study Chair — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen

REFERENCES:
- [Derived] Matzen JS, Krogh CL, Forman JL, Garred P, Moller K, Bache S. Lectin complement pathway initiators after subarachnoid hemorrhage - an observational study. J Neuroinflammation. 2020 Nov 12;17(1):338. doi: 10.1186/s12974-020-01979-y. PMID 33183322
- [Derived] Bache S, Rasmussen R, Rossing M, Laigaard FP, Nielsen FC, Moller K. MicroRNA Changes in Cerebrospinal Fluid After Subarachnoid Hemorrhage. Stroke. 2017 Sep;48(9):2391-2398. doi: 10.1161/STROKEAHA.117.017804. Epub 2017 Aug 2. PMID 28768799